CLINICAL TRIAL: NCT06291194
Title: The Purpose of This Clinical Study is to Prove That the Test Drug (AJU-S56 5%) is Superior to the Control Drug After 24 Weeks of Administration to Patients Who Have Moderate or Severe Dry Eye Syndrome
Brief Title: Efficacy and Safety of AJU-S56 5% in Dry Eye Syndrome Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Collaborators: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22DE30902
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group(AJU-S56 5%) (Experimental): QID(4 times in a day) for 24 Weeks after Randomization
  Interventions: Drug: AJU-S56 5%
- Placebo group(Vehicle) (Placebo Comparator): QID(4 times in a day) for 24 Weeks after Randomization
  Interventions: Drug: Placebo Group(Vehicle)

INTERVENTIONS:
Drug: AJU-S56 5% — After Randomization(Week 0), Participants will be administered with the durg, QID(4 times in a day, and 1 drop per each times) until end of trial(Week 24).
  Other Names: Test Group
  Arms: Test group(AJU-S56 5%)
Drug: Placebo Group(Vehicle) — After Randomization(Week 0), Participants will be administered with the durg, QID(4 times in a day, and 1 drop per each times) until end of trial(Week 24).
  Other Names: Control Group
  Arms: Placebo group(Vehicle)

SUMMARY:
This study is planned to Evaluate the Efficacy and Safety of test drug (AJU-S56 5%) compared to control drug(vehicle) in Patients with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female who over 19 years old
* Moderate to Severe Dry Eye Disease Patients
* Must meet all criteria listed below at least in one eye or both eyes.

  1. TCSS (National eye institute (NEI) scale)≥ 4
  2. Ocular discomfort score (ODS) ≥ 3
  3. Schirmer test(without anesthesia) ≤ 10mm in 5 mins
  4. Tear break-up time ≤ 6 secs
* Written informed consent to participate in the trial

Exclusion Criteria:

* Those who have clinically significant eye disease not related to dry eye syndrome
* Those who have worn contact lenses before 1week Screening visit or have to wear contact lenses or need to wear contact lenses during study period
* Those who have medical history with intraocular surgery 12months before screening visit
* Use of corticosteroid, beta blocker and anticholinergic agent within 4 weeks
* Participation in other studies within 4weeks of screening visit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Total corneal staining score (TCSS) | WEEK 4, 8, 12
  TCSS ≥4 at baseline (Total Max score : 15)

SECONDARY OUTCOMES:
LGCSS | WEEK 4, 8, 12
  Lissamine Green Conjunctival Staining Score(Total score : 0~18)
TFBUT | WEEK 4, 8, 12
  Tear Film Break Up Time

CONTACTS AND LOCATIONS:
Locations (1):
- AJU Pharm Co., Ltd., Seoul, South Korea